CLINICAL TRIAL: NCT06094777
Title: A Phase 1, Multicenter, Open-label, Dose-escalation and Dose-expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HY-0102 Monotherapy in Patients With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Study of HY-0102 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL-0102-02
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor
Keywords: Urothelial carcinoma; Colorectal cancer; Pancreatic cancer; NKG2A; Humanized monoclonal antibody
MeSH Terms: conditions — Carcinoma, Transitional Cell; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HY-0102 (Experimental): Dose Escalation(Standard 3+3 Dose escalation) Cohort 1: 5 mg/kg Q2W HY-0102 ivgtt Duration: 24w,DLT observation period: 28 days.
  Cohort 2: 10 mg/kg Q2W HY-0102 ivgtt Duration: 24w,DLT observation period: 28 days.
  Cohort 3: 15 mg/kg Q2W HY-0102 ivgtt Duration: 24w,DLT observation period: 28 days.
  Dose Expansion Within the MTD and sub-MTD dose groups, select 1-2 doses for dose expansion, including approximately 30-40 cases of tumor types that have demonstrated preliminary efficacy in the early escalation phase. Conduct safety, tolerability, and preliminary anti-tumor efficacy evaluations to provide a basis for the recommended phase II clinical dose (RP2D). PK studies will be conducted on 12 subjects in each dose group, including dose escalation trial cases.
  Interventions: Drug: HY-0102

INTERVENTIONS:
Drug: HY-0102 — Multiple dose cohorts, 60 minute IV infusion, every two weeks, 28 days as a cycle

SUMMARY:
This is a phase 1 open label multicenter study to evaluate the maximum tolerance, safety, tolerance and PK of HY-0102 administered intravenously (IV) once every two weeks in patients with advanced solid tumors, so as to confirm the recommended phase 2 dose of HY-0102 and obtain the preliminary efficacy information of patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase I trial to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of HY-0102 administered intravenously (IV) once every two weeks in adult patients with locally advanced/metastatic malignant solid tumors (urothelial carcinoma, colorectal and pancreatic cancers, etc).

Three dosing cohorts are planned with the doses of 5, 10 and 15 mg/kg. The study will apply a standard 3+3 dose escalation design in dose escalation.Dose expansion will enroll approximately 30-40 cases of tumor types that have demonstrated preliminary efficacy in the early escalation phase.

The number of enrolled patients is estimated to be up to 50. The dose limiting toxicity evaluation period will be the first 28 days (Cycle 1) and subsequent cycles will be 4 weeks in duration. Patients will receive the investigational drug on Day 1 of cycle 1 followed by 28 days of observation. HY-0102 will be administered IV once every two weeks for Cycle 2 and beyond.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet the following criteria to be considered for inclusion in the study:

1. Demonstrated willingness to voluntarily provide a signed informed consent document.
2. Male or female individuals aged ≥18 years.
3. Advanced malignant solid tumor patients who have experienced treatment failure using established therapeutic methods, have no viable standard treatment options available, or are unable to tolerate standard therapy. (Preference will be given to patients with urothelial carcinoma, colorectal cancer, and pancreatic cancer)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Anticipated minimum survival duration of 3 months.
6. Measurable or evaluable lesions detected by CT/MRI scans; participants in the dose expansion phase must have quantifiable lesions according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). Measurable lesions may also include those located in previously irradiated (or subjected to other local therapy) areas, demonstrating evident progression as confirmed by post-radiation therapy imaging.
7. Participants must meet the following laboratory criteria with adequate organ and bone marrow function prior to enrollment:

1) Bone marrow reserve (no blood transfusion or blood product administration within 14 days preceding the first dose, absence of the use of G-CSF or other hematopoietic growth factors for correction): Absolute neutrophil count (ANC) ≥1.5×109/L, white blood cell count (WBC) ≥3.0×109/L, hemoglobin (HB) ≥90 g/L, platelet count (PLT) ≥100×109/L (patients with hepatocellular carcinoma (HCC) may have PLT ≥75×109/L); 2) Liver function: Alanine transaminase (ALT) ≤3×upper limit of normal (ULN), aspartate transaminase (AST) ≤3×ULN, alkaline phosphatase (ALP) ≤2.5×ULN, total bilirubin (TBIL) ≤1.5×ULN (patients with known Gilbert's syndrome and serum bilirubin level ≤3 times ULN can be included), liver metastasis patients: ALT ≤5×ULN, AST ≤5×ULN, ALP ≤5×ULN); 3) Renal function: Creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min calculated using the Cockcroft-Gault formula; 4) Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5×ULN (for patients not on anticoagulant therapy, inclusion can be determined by the investigator); 8. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to utilize highly effective contraception methods throughout the treatment period (with a failure rate of less than 1% when used correctly and consistently). Participants receiving HY-0102 treatment should continue contraception for 6 months following the final dose administration. Acceptable contraceptive methods include combined hormonal contraception (including estrogen or progestogen), progestogen-only pills primarily inhibiting ovulation when combined with another barrier method (typically containing a spermicide), intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomy, and sexual abstinence.

1. Considering potential interactions between the investigational drug and oral contraceptives, oral contraceptives should always be combined with alternative contraceptive methods. This requirement also applies to male participants with partners of childbearing potential, who must utilize condoms.
2. Non-menopausal (non-treatment-related amenorrhea for ≥12 months) or non-sterilized female participants must obtain a negative serum pregnancy test result within 7 days prior to initiating the study drug.
3. Women who have undergone tubal ligation or hysterectomy are exempt from contraception requirements.

9. Participants must have sufficiently recovered from all acute toxicities resulting from previous treatment (recovery to Grade 1 or below), excluding alopecia, hyperpigmentation, peripheral neuropathy recovered to <CTCAE Grade 2, and long-term toxicities caused by radiation therapy, at the discretion of the investigator.

Exclusion Criteria:

-

Participants will be excluded if they meet any of the following criteria:

1. Allergies or hypersensitivity to any component of the investigational product.
2. Severe or uncontrolled cardiac diseases, congestive heart failure graded as III or IV according to the New York Heart Association (NYHA), unstable angina that cannot be controlled with medication, history of myocardial infarction within the previous 6 months, or severe arrhythmias requiring medication (excluding atrial fibrillation or paroxysmal supraventricular tachycardia).
3. Active seizures requiring antiepileptic drugs, recent (< 6 months) cerebrovascular accidents or transient ischemic attacks.
4. Symptomatic brain metastases or untreated brain metastases meeting at least one of the following criteria:

   1. Requires the use of corticosteroids or dehydration therapy (excluding antiepileptic drugs after surgery or radiation therapy);
   2. Presents with clinically significant symptoms;
   3. Tumor stability lasting less than 4 weeks after radiation therapy or surgery.
5. Requires oxygen therapy for daily activities; asthma requiring medical intervention with bronchodilators.
6. Peripheral neuropathy of Grade ≥2.
7. Received any chemotherapy, hormonal therapy, radiation therapy, immunotherapy, or biological therapy within 4 weeks prior to the first dose of the investigational treatment, or within 5 half-lives of the previous treatment, whichever is shorter. The following exceptions are allowed:

   1. Local topical or inhaled corticosteroids;
   2. Short-term (≤7 days) use of corticosteroids for prophylaxis or treatment of non-autoimmune allergy disorders;
   3. Local palliative radiation therapy for bone metastases.
8. Underwent major surgery within 4 weeks prior to enrollment or has not fully recovered from previous surgery (definition of major surgery according to the "Management Measures for Clinical Application of Medical Technologies" implemented on May 1, 2009) or anticipates significant surgery within 28 days during the study.
9. Participants with autoimmune diseases or history of autoimmune diseases, including but not limited to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis (participants with resolved childhood asthma or vitiligo without any intervention in adulthood may be included).
10. Active viral, bacterial, fungal, or other infections requiring systemic treatment (excluding onychomycosis).
11. Active hepatitis B (positive for hepatitis B surface antigen and/or positive for hepatitis B core antibody with HBV-DNA ≥10^4 copies/mL or ≥2000 IU/mL), active hepatitis C (positive for hepatitis C virus antibodies and/or positive for HCV-RNA), or positive HIV test.
12. Severe infection within 4 weeks prior to first dose administration or active infection requiring oral or intravenous antibiotic treatment within the past 2 weeks as determined by the investigator.
13. Participants with severe concurrent chronic or acute diseases (e.g., cardiovascular or pulmonary diseases, liver diseases, or diseases that the investigator considers as high risk for experimental drug treatment).
14. History of any malignancy within the past 3 years, with the exception of cured basal cell carcinoma, squamous cell carcinoma of the skin, thyroid cancer, cervical carcinoma in situ, or primary lung adenocarcinoma.
15. Vaccination with a live attenuated vaccine within 4 weeks prior to the first dose of study medication or planned administration during the study period.
16. Pregnancy or breastfeeding.
17. Left ventricular ejection fraction (LVEF) <45% as shown on transthoracic echocardiography (ECHO) or multiple gated acquisition (MUGA) scanning.
18. Fridericia-corrected QT interval (QTcF) >480 milliseconds.
19. The investigator believes that there are clinically significant conditions or factors that may affect compliance with the treatment regimen, the participant's ability to provide informed consent, or suitability for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of drug limited toxicities (DLTs) | From Time of First dose through DLT observation period, 28 days
  To assess by the occurrence of Drug Limited Toxicities (DLTs)
Incidence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs) | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess by the occurrence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs)
Number of patients with changes in laboratory parameters from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102
Number of patients with changes in electrocariogram (ECG) from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102
Number of participants with changes in clinically significant vital sign from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102

SECONDARY OUTCOMES:
ORR (confirmed complete or partial response) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 12 months
  The overall response rate (ORR) will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1
DCR (confirmed response or stable disease lasting for at least 6 months) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 12 months
  According to the RECIST v1.1 to assess anti-tumor activity of HY-0102
Duration of Response (DoR) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 12 months
  According to the RECIST v1.1 to assess anti-tumor activity of HY-0102
Progression Free Survival (PFS) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 6 months
  According to the RECIST v1.1 to assess anti-tumor activity of HY-0102
Cmax (Maximum observed serum concentration) of HY-0102 | From first dose through 30days(±7) days after the last dose of study medication
  Cmax of HY-0102 is observed directly from data
Ctrough (Trough observed serum concentration) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  Ctrough of HY-0102 was observed directly from data.
Tmax(Time to maximum plasma concentration) | From first dose through 30(±7) days after the last dose of study medication
  Tmax of HY-0102 was observed directly from data as time of Cmax.
AUC(0-T) [Area under the concentration-time curve from time zero to the last quantifiable concentration] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUClast of HY-0102 was determined by linear/log trapezoidal method.
AUC(tau) [Area under the concentration-time curve in one dosing interval] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUCtau of HY-0102 was determined using linear/log trapezoidal method.
AUC(inf) [Area under the concentration-time curve from time zero to infinity and the extrapolated area] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUCinf = AUClast + (Clast*/kel), where Clast* is the estimated concentration at the time of the last measurable concentration and kel is the terminal phase rate constant calculated as the absolute value of the slope of a linear regression during the terminal phase of the natural log-transformed concentration time profile.
T1/2 (Elimination half life) of HY-0102 | From first dose through 30 days (+/- 7 days) after the last dose of study medication
  T1/2 of HY-0102 was observed directly from data.
Anti-drug Antibody (ADA) | From first dose through 30(±7) days after the last dose of study medication
  To assess the immunogenicity of HY-0102

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No